CLINICAL TRIAL: NCT00750672
Title: Follow-up After Primary Therapy for Endometrial Cancer; Implementation of a Cancer Care Ontario Guideline: A Pilot Evaluation Study.
Brief Title: Follow-up Care After Treatment for Endometrial Cancer
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Ottawa Regional Cancer Centre (Other)
Responsible Party: Sponsor
Other Study IDs: OHRI 2008-361; 2008361-01H for OHREB
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Endometrial Neoplasm
Keywords: Endometrial neoplasia; Follow-up care; survivorship; Primary care provider
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purposes of this study are to examine the needs (symptoms, support, information) and satisfaction of women during follow-up in the community after completing treatment for endometrial cancer. This information will be collected from the perspective of the women themselves, their primary care providers (family physician or gynecologist) and the health care providers (oncologist, nurses, social worker, psychologist) at the cancer centre.

DETAILED DESCRIPTION:
Research Question How has this transfer in follow-up care impacted performance indicators?

* Volume of follow-up care transferred
* Percentage of women, who have required a re-entry consultation
* Fiscal implication of this transfer of follow-up care

Patient stakeholders:

* What are women's perceptions of the transition of follow-up care?
* What are women's supportive care needs during the transition of follow-up care and ongoing needs?

Primary Care Practitioner stakeholders:

* What are the primary care practitioners' perceptions of the process of transition of follow-up care?
* What are the primary care practitioners' educational needs?
* What are the primary care practitioners' perceptions of the process of re-entry for in women with suspected recurrence?

Tertiary Centre: Health care providers stakeholders

o What are the perceptions of tertiary health care providers about the transition of follow-up care?

ELIGIBILITY:
Inclusion Criteria:

* Participants- women diagnosed with endometrial cancer:

  * 18 years of age or older.
  * speak English or French
  * who have been treated (surgery and/or radiation therapy) at TOH.
  * who have been discharged from follow-up in the cancer centre in the past 6 months.
* Participants-primary care provider practitioner:

  * providing follow-up care to at least one woman with endometrial cancer
* Participants- health care providers at the tertiary centre :

  * physicians, nurses or allied health care providers whose primary responsibility are to provide care to women with gynecological cancer.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will employ a convenience sample of women with endometrial cancer treated at the Ottawa Hospital Cancer Centre who have been discharged from follow-up after September 2005. Women will be identified from the Cancer Centre health records. The primary care providers will also be identified by health records as provided by the endometrial cancer patient when they registered with the TOHCC.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-08; Primary Completion 2009-09 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Qualitative description of participants perception | after 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada